CLINICAL TRIAL: NCT04251286
Title: Screening and Follow-up Study of Neonatal Jaundice Based on Mobile Network：A Multicentrd, Prospective, Open, Clinical Study
Brief Title: Screening and Follow-up Study of Neonatal Jaundice Based on Mobile Network
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: Xuzhou Maternity and Child Health Care Hospital (Other); Jiangsu Women and Children Health Hospital (Unknown); Changzhou Maternal and Child Care Hospital (Other); Lianyungang Maternity and Child Health Care Hospital (Unknown); Affiliated Hospital of Jiangsu University (Other); Suqian First Hospital (Other); Jiangyin People's Hospital (Other); Nantong Maternity and Child Health Care Hospital (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Taizhou People's Hospital (Unknown); Yangzhou Maternity and Child Health Care Hospital (Unknown); Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Principal Investigator of Nan Jing Maternity and Child Health Care Hospital, Nanjing Medical University
Other Study IDs: NMU-FY2018-54
Record Dates: First submitted 2020-01-16; First posted 2020-01-31 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; screening; follow-up
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At least 13 hospitals in China will participate in the study, which aims to clarify the natural history of jaundice in Chinese healthy newborns，and decrease the incidence of severe hyperbilirubinemia and acute bilirubin encephalopathy and even kernicterus. The study is an open project, and the investigators welcome institutions fulfilling the specified requirements to join the study during the recruitment phase.

DETAILED DESCRIPTION:
This is a prospective cohort study of healthy term and near-term infants. The mobile network screening and follow-up of neonatal jaundice consists of two parts, one is the screening and follow-up program for healthy neonatal jaundice by using on parents' mobile phones, the other is the online registry of severe hyperbilirubinemia. Firstly，the TCB values of healthy term and near-term infants in delivery institutions will be prospectively recorded and followed up until jaundice subsided by using screening and follow-up program, so as to clarify the natural history of jaundice of healthy newborns in China. Secondly, by establishing an online registry for severe hyperbilirubinemia and "Follow up of jaundice" on Wechat applet, the investigators will find the specific problems of jaundice management in infants with severe hyperbilirubinemia. Lastly, through the follow-up of severe hyperbilirubinemia cases, the investigators will have a better understanding of their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Term or near-term neonates with gestational age ≥35w and birth weight ≥2000g.

Exclusion Criteria:

* Biliary atresia, serious genetic and metabolic diseases, family history of epilepsy, and so on.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For the research on the natural history of jaundice via mobile network, the selected population is healthy newborns with gestational age ≥35 weeks and weight ≥2000g, and those without phototherapy or hospital intervention. For the study of the online registry for severe hyperbilirubinemia, the study population is gestational age ≥35 weeks, weight ≥2000g, only hospitalized for jaundice, and the serum total bilirubin reached the threshold of exchange transfusion (≤3 days) or the serum total bilirubin ≥20mg / dl (>3 days).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
To record the TCB values of Chinese newborns within 28 days after birth. | 12 months
  Transcutaneous bilirubin (TcB) values will be recorded so as to establish transcutaneous bilirubin nomogram in healthy Chinese term and late-preterm infants at <28 days of age.
The comprehensive prognosis of infants | 60 months
  To investigate the comprehensive prognosis of infants with severe hyperbilirubinemia at the corrected age of 2 years in a real-world setting in Jiangsu Province.

SECONDARY OUTCOMES:
Risk factors of extreme hyperbilirubinemia | 36 months
  Extreme hyperbilirubinemia:total serum bilirubin more than 25mg/dL.
The incidence of neurological sequelae. | 60 months
  To assess the clinical outcome at 2 years of corrected age in cases treated with and without exchange transfusion when TSB is at a level of the threshold
The completion rate of each jaundice management measure for severe hyperbilirubinemia cases. | 36 months
  To calculate the completion rate of each jaundice management measure for severe hyperbilirubinemia cases, whose total serum bilirubin are more than 20mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Han Shuping, PHD, Study Director — Nanjing Maternity and Child Health Care Hospital; Yu Zhangbin, PHD, Study Director — Nanjing Maternity and Child Health Care Hospital; Deng Xiaoyi, MD, Principal Investigator — Xuzhou Maternity and Child Health Care Hospital; Hu Yuhua, PHD, Principal Investigator — Jiangsu Women and Children Health Hospital; Wang Jinxiu, PHD, Principal Investigator — Changzhou Maternal and Child Care Hospital; Li Qianqian, MD, Principal Investigator — Xuzhou Maternity and Child Health Care Hospital; Gao Yan, MD, Principal Investigator — Lianyungang Maternity and Child Health Care Hospital; Lu Hongyan, MD, Principal Investigator — Affiliated Hospital of Jiangsu University; Zhang Jia, MD, Principal Investigator — Suqian First Hospital; Wan Jun, MD, Principal Investigator — Jiangyin People's Hospital; Li Shuangshuang, MD, Principal Investigator — Nantong Maternity and Child Health Care Hospital; Wu Mingfu, MD, Principal Investigator — Yangzhou University; Wu Xinping, MD, Principal Investigator — Yangzhou Maternity and Child Health Care Hospital; Wang Jun, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Xue Mei, MD, Principal Investigator — Taizhou People's Hospital
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The study is an open project, and the collected data and information will be provided to all participating centers after review by the data management committee. Anyone interested in this research can contact us directly.
Supporting Information: Study Protocol
Time Frame: The Study Protocol will be shared after the publication until the end of the study.
Access Criteria: All participating centres

REFERENCES:
- [Derived] Li Q, Deng X, Yan J, Sun X, Dong X, Chen X, Han S, Huo J, Yu Z. Neonatal Severe Hyperbilirubinemia Online Registry in Jiangsu Province: protocol for a multicentre, prospective, open, observational cohort study. BMJ Open. 2021 Feb 5;11(2):e040797. doi: 10.1136/bmjopen-2020-040797. PMID 33550236